CLINICAL TRIAL: NCT02283203
Title: A Double-blind, Randomized, Placebo-controlled Phase IV Clinical Study of the Efficacy and Safety of a New Formulation of Paracetamol for the Management of Fever of Infectious Origin
Brief Title: A New Formulation of Intravenous Paracetamol for Fever Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Uni-Pharma Kleon Tsetis Pharmaceutical Laboratories S.A. (Industry)
Collaborators: Attikon Hospital (Other); University Hospital of Patras (Other); University Hospital of Crete (Other); Thriasio General Hospital of Elefsina (Other); General Hospital Of Thessaloniki Ippokratio (Other); General Hospital of Chalkida (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: APOTEL-02
Record Dates: First submitted 2014-10-19; First posted 2014-11-05 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Fever
Keywords: Paracetamol; Management of fever; Infections
MeSH Terms: conditions — Fever; Infections | interventions — Water; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- APOTEL max (Active Comparator): Active drug; water for injection at a volume of 100ml with added 1g of paracetamol and inactive ingredients (ΑPOTEL max®), infused within 15 minutes. Available in 100ml bags.
  Interventions: Drug: APOTEL max
- Placebo (Placebo Comparator): Placebo; water for injection at a volume of 100ml with added inactive ingredients, infused within 15 minutes. Available in 100ml bags.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: APOTEL max — The study drug is provided in a form of bag with 100ml final volume and it is directly connected to the infusion device that leads to a catheter already cannulated in one antecubital vein.
  Other Names: Paracetamol solution for infusion, 1gram per 100ml bag
  Arms: APOTEL max
Drug: Placebo — Placebo is provided in a form of bag with 100ml final volume and it is directly connected to the infusion device that leads to a catheter already cannulated in one antecubital vein. Placebo contains water for injection and inactive vehicles.
  Other Names: Water for injection and vehicles
  Arms: Placebo

SUMMARY:
The efficacy of intravenous paracetamol has never been compared with other drugs for the management of fever due to infections. Available data come from clinical studies conducted in healthy volunteers subject to experimental endotoxemia. The present study compares the efficacy of the new ΑPOTEL Μax® formulation versus placebo for the management of fever of infectious origin.

DETAILED DESCRIPTION:
A new formulation of paracetamol for intravenous administration has been manufactured in Greece by the industry Uni-Pharma (ΑPOTEL Μax®). According to this new formulation, 1g of paracetamol is provided as a flask diluted into 100ml volume with the possibility of immediate connection with the infusion device of the patient. This formulation provides the advantage of a dilution ready-to-use which equals considerable financial benefit; nursing staff is not pre-occupied with the preparation of dilutions and the amount of consumables required for the preparation of this dilution is significantly decreased. Taking into consideration that the antipyretic effect of intravenous paracetamol has never been studied compared with other agents in patients and available data come from studies in volunteers with experimental endotoxemia, the present study compares the efficacy of the new ΑPOTEL Μax® formulation versus placebo for the management of fever of infectious origin (fever due to infection of the upper respiratory tract, of the lower respiratory tract, acute pyelonephritis or of the skin and soft tissues).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent by the patient
2. Patient of either gender
3. Age equal to or greater than 18 years old
4. Fever onset less than 24 hours
5. Body temperature greater than or equal to 38.50C.
6. Infection of the upper respiratory tract or of the lower respiratory tract or acute pyelonephritis or infection of the skin and soft tissues that can explain fever onset.

Exclusion Criteria:

1. Age below 18 years old
2. Denial for written consent
3. Intake of paracetamol for any reason either orally or intravenously or intramuscularly the last 12 hours
4. Intake of any non-steroidal anti-inflammatory drug the last 8 hours
5. Intake of any steroidal anti-inflammatory drug the last 12 hours
6. History of liver cirrhosis
7. Serum creatinine greater than 3 mg/dl
8. Aspartate aminotransferase more than 3 times greater than the upper normal limit for the hospital lab
9. Known allergy to non-steroidal anti-inflammatory drugs or to paracetamol
10. Pregnancy or lactation
11. Active bleeding of the upper or the lower gastrointestinal tract
12. Thrombocytopenia defined as any absolute platelet count below 50000/mm3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Body temperature as a measure of to compare the efficacy of intravenously administered ΑPOTEL Μax® over placebo for the achievement of defervescence. | 3 hours
  The comparative efficacy of intravenously administered ΑPOTEL Μax® over placebo for the achievement of defervescence; defervescence is defined as any body temperature equal to or lower than 37.1 degC.

SECONDARY OUTCOMES:
Need for the administration of rescue drug. | 30 hours
  The comparison between the two study groups on the frequency and time to administration of rescue drug.
Comparison of defervescence with the rescue drug in the paracetamol arm with the placebo arm | 30 hours
  The correlation between defervescence with the rescue drug with the efficacy of the initially administered type of study drug (placebo over active drug).
Correlation between serum concentrations of free active paracetamol and metabolites with the clinical efficacy of paracetamol | 30 hours
  The correlation between the achievement of defervescence and the concentrations of free active paracetamol and its metabolites in the serum of the patients.
The administration of other antipyretics by the attending physicians after rescue drug in each study group | 30 hours
  The correlation between achievement of defervescence with the rescue drug and the need of further administration of other drugs as antipyretics at the discretion of the attending physicians.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Boumpas, MD, PhD, Principal Investigator — Attikon Hospital; Charalambos Gogos, MD, PhD, Principal Investigator — University Hospital of Patras; George Samonis, MD, PhD, Principal Investigator — University Hospital of Crete; Styliani Sympardi, MD, Principal Investigator — Thriasio General Hospital of Elefsina; Asterios Karagiannis, MD, PhD, Principal Investigator — University Hospital of Thessaloniki Hippokrateion; Nikolaos Tsokos, MD, Principal Investigator — General Hospital of Halkida
Locations (6):
- Greece (6):
  - General Hospital of Chalkida, Chalcis
  - Attikon Hospital, Haidari/Athens
  - University Hospital of Crete, Heraklion
  - Thriasion Elefsis General Hospital, Magoula Attikis
  - University Hospital of Patras, Rion/Patras
  - General Hospital Of Thessaloniki Ippokratio, Thessaloniki

REFERENCES:
- [Background] Giamarellos-Bourboulis EJ, Spyridaki A, Savva A, Georgitsi M, Tsaganos T, Mouktaroudi M, Raftogiannis M, Antonopoulou A, Papaziogas V, Baziaka F, Sereti K, Christopoulos P, Marioli A, Kanni T, Maravitsa P, Pantelidou I, Leventogiannis K, Tsiaoussis P, Lymberopoulou K, Koutelidakis IM. Intravenous paracetamol as an antipyretic and analgesic medication: the significance of drug metabolism. J Pharmacol Sci. 2014;124(2):144-52. doi: 10.1254/jphs.13133fp. Epub 2014 Jan 30. PMID 24553403